CLINICAL TRIAL: NCT01347086
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses (400mg, 800mg, 1200mg) of BI 207127 NA in Healthy Male Asian Volunteers and Single Oral Dose (1200 mg) of BI 207127 NA in Healthy Male Caucasian Volunteers (Randomised, Double-blind, Placebo-controlled Within Dose Group)
Brief Title: Single Rising Dose Study of BI 207127 NA in Healthy Male Asian Volunteers and Single Dose Study of BI 207127 NA in Healthy Male Caucasian Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1241.8
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Healthy

ARMS (6):
- BI 207127 NA (low dose) (Experimental): Single dose of BI 207127 NA
  Interventions: Drug: BI 207127 NA (low dose)
- Matching placebo (low dose) (Placebo Comparator): Single dose of matching placebo
  Interventions: Drug: Matching placebo (low dose)
- BI 207127 NA (medium dose) (Experimental): Single dose of BI 207127 NA
  Interventions: Drug: BI 207127 NA (medium dose)
- Matching placebo (medium dose) (Placebo Comparator): Single dose of matching placebo
  Interventions: Drug: Matching placebo (medium dose)
- BI 207127 NA (high dose) (Experimental): Single dose of BI 207127 NA
  Interventions: Drug: BI 207127 NA (high dose)
- Matching placebo (high dose) (Placebo Comparator): Single dose of matching placebo
  Interventions: Drug: Matching placebo (high dose)

INTERVENTIONS:
Drug: Matching placebo (low dose) — single dose of matching placebo
  Arms: Matching placebo (low dose)
Drug: BI 207127 NA (medium dose) — Single does of BI 207127 NA
  Arms: BI 207127 NA (medium dose)
Drug: BI 207127 NA (low dose) — single dose of BI 207127 NA
  Arms: BI 207127 NA (low dose)
Drug: Matching placebo (medium dose) — Single dose of matching placebo
  Arms: Matching placebo (medium dose)
Drug: BI 207127 NA (high dose) — Single dose of BI 207127 NA
  Arms: BI 207127 NA (high dose)
Drug: Matching placebo (high dose) — Single dose of matching placebo
  Arms: Matching placebo (high dose)

SUMMARY:
The aim of the study is to evaluate safety, tolerability and pharmacokinetics in Asian and Caucasian healthy male volunteers administered BI 207127 NA.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male volunteers
2. Chinese ethnicity or Japanese ethnicity or Caucasian
3. Body Mass Index (BMI) = 18.5 and BMI =25 kg/m2 for Japanese and Chinese, BMI =18.5 and BMI = 29.9 kg/m2 for Caucasians

Exclusion criteria:

1. Any finding of the medical examination (including Blood pressure(BP), Pulse rate (PR) and Electrocardiogram (ECG)) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1241.8.8201 Boehringer Ingelheim Investigational Site, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 subjects were included (27 Chinese, 25 Japanese, and 8 Caucasian subjects). 24 Japanese and 24 Chinese subjects were randomised to 1 of 3 (rising) dose groups and received single oral doses of either 400mg, 800mg, or 1200mg of BI 207127 NA or of the respective placebo. Caucasian subjects were randomised to 1200 mg BI 207127 NA or placebo.
Pre-assignment Details: The decision to proceed to the next higher dose group was based upon the safety of the preceding dose group. Caucasian subjects were randomised to receive either placebo or 1200 mg BI 207127 NA; this dose group could be started independently from the results of dose escalation in the Asian subjects.
Groups:
- Placebo (Caucasian Subjects): Caucasian subjects who received matching placebo.
  Oral with 240 mL of water in fed condition.
- 1200 mg Deleobuvir (Caucasian Subjects): Caucasian subjects who received 1200 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
- Placebo (Japanese Subjects): Japanese subjects who received matching placebo.
  Oral with 240 mL of water in fed condition.
- 400 mg Deleobuvir (Japanese Subjects): Japanese subjects who received 400 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
- 800 mg Deleobuvir (Japanese Subjects): Japanese subjects who received 800 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
- 1200mg Deleobuvir (Japanese Subjects): Japanese subjects who received 1200 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
- Placebo (Chinese Subjects): Chinese subjects who received matching placebo.
  Oral with 240 mL of water in fed condition.
- 400 mg Deleobuvir (Chinese Subjects): Chinese subjects who received 400 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
- 800 mg Deleobuvir (Chinese Subjects): Chinese subjects who received 800 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
- 1200 mg Deleobuvir (Chinese Subjects): Chinese subjects who received 1200 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
Period: Overall Study
Arm/Group | Placebo (Caucasian Subjects) | 1200 mg Deleobuvir (Caucasian Subjects) | Placebo (Japanese Subjects) | 400 mg Deleobuvir (Japanese Subjects) | 800 mg Deleobuvir (Japanese Subjects) | 1200mg Deleobuvir (Japanese Subjects) | Placebo (Chinese Subjects) | 400 mg Deleobuvir (Chinese Subjects) | 800 mg Deleobuvir (Chinese Subjects) | 1200 mg Deleobuvir (Chinese Subjects)
Started | 2 | 6 | 7 (2 participants were treated together with each dose level of Deleobuvir. 1 subject was not treated.) | 6 | 6 | 6 | 7 (2 participants treated together with each dose level of Deleobuvir. 1 subject was not treated.) | 7 (One subject was not treated.) | 6 | 7 (One subject was not treated.)
Completed | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — failed screening visit | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The treated set (full analysis set according to ICH-E9): all subjects who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1200 mg Deleobuvir (Caucasian Subjects) | Placebo (Caucasian Subjects) | 400 mg Deleobuvir (Japanese Subjects) | 800 mg Deleobuvir (Japanese Subjects) | 1200mg Deleobuvir (Japanese Subjects) | Placebo (Japanese Subjects) | 400 mg Deleobuvir (Chinese Subjects) | 800 mg Deleobuvir (Chinese Subjects) | 1200 mg Deleobuvir (Chinese Subjects) | Placebo (Chinese Subjects) | Total
Number analyzed (Participants) | 6 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (7.0) | 31.0 (8.5) | 28.8 (7.0) | 28.2 (4.6) | 23.7 (3.6) | 29.2 (7.1) | 24.7 (2.1) | 26.0 (3.9) | 23.7 (2.3) | 23.0 (2.1) | 26.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drug Related Adverse Events
Description: Number of subjects with investigator-defined drug-related adverse events (AEs). Tolerability assessment endpoint.
  The investigator assessed the possible causal relationship between all AEs and the investigational drug, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, and confounding factors such as concomitant medication, concomitant diseases, and relevant history.
Time Frame: From first administration of study drug (drug related AEs) until 14 days after end of trial visit, upto 17 days.
Population: Treated set (full analysis set according to the International Conference on Harmonization (ICH) E9 guideline): all subjects who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Measure: Number; unit: Participants
Arm/Group | 1200 mg Deleobuvir (Caucasian Subjects) | Placebo (Caucasian Subjects) | 400 mg Deleobuvir (Japanese Subjects) | 800 mg Deleobuvir (Japanese Subjects) | 1200mg Deleobuvir (Japanese Subjects) | Placebo (Japanese Subjects) | 400 mg Deleobuvir (Chinese Subjects) | 800 mg Deleobuvir (Chinese Subjects) | 1200 mg Deleobuvir (Chinese Subjects) | Placebo (Chinese Subjects)
Number analyzed (Participants) | 6 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 5 | 1 | 0 | 0 | 5 | 2 | 1 | 2 | 4 | 2

2. Primary Outcome: Number of Subjects With Adverse Events as Determined by Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinanalysis and ECG
Description: Clinical relevant abnormalities for vital signs, blood chemistry, haematology, urinanalysis and ECG. Tolerability assessment endpoint.
  New abnormal findings or worsening of baseline conditions were reported as adverse events. Adverse events were assessed through the entire trial, from signing the informed consent (within 21 days before drug administration) onwards through the observational phase until the end-of-trial-examination (within 14 days after last trial procedure).
Time Frame: From signing the informed consent (within 21 days before drug administration) until 14 days after end of trial visit, upto 38 days.
Population: The treated set.
Measure: Number; unit: participants
Arm/Group | 1200 mg Deleobuvir (Caucasian Subjects) | Placebo (Caucasian Subjects) | 400 mg Deleobuvir (Japanese Subjects) | 800 mg Deleobuvir (Japanese Subjects) | 1200mg Deleobuvir (Japanese Subjects) | Placebo (Japanese Subjects) | 400 mg Deleobuvir (Chinese Subjects) | 800 mg Deleobuvir (Chinese Subjects) | 1200 mg Deleobuvir (Chinese Subjects) | Placebo (Chinese Subjects)
Number analyzed (Participants) | 6 | 2 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: AUC0-∞ of Deleobuvir
Description: Area under the concentration-time curve of the analyte in plasma (Deleobuvir) over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: -2:00, 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 10:00, 12:00, 24:00, 36:00, 48:00 h (hours) after drug administration
Population: The pharmacokinetic (PK) analysis set: all evaluable subjects of the treated set who provided at least 1 observation for at least 1 PK endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol*h/L
Groups:
- Caucasian 1200 mg: Caucasian subjects who received a single dose of 1200 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
- Japanese 400 mg: Japanese subjects who received a single dose of 400 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
- Japanese 800 mg: Japanese subjects who received a single dose of 800 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
- Japanese 1200 mg: Japanese subjects who received a single dose of 1200 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
- Chinese 400 mg: Chinese subjects who received a single dose of 400 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
- Chinese 800 mg: Chinese subjects who received a single dose of 800 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
- Chinese 1200 mg: Chinese subjects who received a single dose of 1200 mg Deleobuvir.
  Oral with 240 mL of water in fed condition.
Arm/Group | Caucasian 1200 mg | Japanese 400 mg | Japanese 800 mg | Japanese 1200 mg | Chinese 400 mg | Chinese 800 mg | Chinese 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6
µmol*h/L | 61.2 (45.5) | 14.0 (56.1) | 31.4 (52.3) | 48.2 (39.1) | 8.7 (78.7) | 42.6 (28.2) | 72.0 (55.9)

4. Secondary Outcome: Tmax of Deleobuvir
Description: Time from dosing to the maximum measured concentration of the analyte in plasma (Deleobuvir).
Time Frame: -2:00, 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 8:00, 10:00, 12:00, 24:00, 36:00, 48:00 h after drug administration
Population: The PK analysis set.
Measure: Median (Full Range); unit: h
Arm/Group | Caucasian 1200 mg | Japanese 400 mg | Japanese 800 mg | Japanese 1200 mg | Chinese 400 mg | Chinese 800 mg | Chinese 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6
h | 6.01 [5.00 to 8.00] | 4.51 [4.00 to 6.02] | 5.50 [4.00 to 6.00] | 5.00 [4.00 to 6.00] | 4.50 [2.50 to 5.00] | 5.00 [4.00 to 6.00] | 5.50 [4.00 to 6.00]

5. Secondary Outcome: Cmax of Deleobuvir
Description: Maximum measured concentration of the analyte in plasma (Deleobuvir).
Time Frame: as for outcome 4
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol/L
Arm/Group | Caucasian 1200 mg | Japanese 400 mg | Japanese 800 mg | Japanese 1200 mg | Chinese 400 mg | Chinese 800 mg | Chinese 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6
µmol/L | 11.8 (42.0) | 3.2 (63.9) | 6.41 (47.4) | 8.26 (37.7) | 2.32 (75.5) | 8.89 (24.1) | 12.9 (51.3)

6. Secondary Outcome: AUC0-∞ of BI 208333 (Metabolite of Deleobuvir)
Description: Area under the concentration-time curve of the analyte in plasma (BI 208333) over the time interval from 0 extrapolated to infinity. The descriptive statistics of the arms "Japanese 400mg", "Japanese 800mg" and "Chinese 400mg" cannot be determined. The reason was that there were too few data to derive a terminal elimination rate constant (slope) to calculate AUC0-∞.
Time Frame: as for outcome 4
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol*h/L
Arm/Group | Caucasian 1200 mg | Japanese 1200 mg | Chinese 800 mg | Chinese 1200 mg
Number analyzed (Participants) | 6 | 5 | 5 | 5
µmol*h/L | 12.7 (54.6) | 10.1 (54.2) | 5.97 (23.9) | 9.01 (186.0)

7. Secondary Outcome: Tmax of BI 208333 (Metabolite of Deleobuvir)
Description: Time from dosing to the maximum measured concentration of the analyte in plasma (BI 208333) .
Time Frame: as for outcome 4
Population: The PK analysis set.
Measure: Median (Full Range); unit: h
Arm/Group | Caucasian 1200 mg | Japanese 400 mg | Japanese 800 mg | Japanese 1200 mg | Chinese 400 mg | Chinese 800 mg | Chinese 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6
h | 6.00 [5.00 to 8.00] | 6.00 [4.00 to 8.00] | 6.00 [4.00 to 8.00] | 6.00 [5.00 to 6.00] | 5.01 [3.97 to 6.00] | 6.00 [5.00 to 8.00] | 6.00 [4.00 to 10.00]

8. Secondary Outcome: Cmax of BI 208333 (Metabolite of Deleobuvir)
Description: Maximum measured concentration of the analyte in plasma (BI 208333).
Time Frame: as for outcome 4
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol/L
Arm/Group | Caucasian 1200 mg | Japanese 400 mg | Japanese 800 mg | Japanese 1200 mg | Chinese 400 mg | Chinese 800 mg | Chinese 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6
µmol/L | 1.82 (42.8) | 0.59 (43.6) | 0.92 (54.2) | 1.32 (55.0) | 0.58 (26.8) | 0.86 (38.9) | 1.19 (104.0)

9. Secondary Outcome: AUC0-∞ of CD 6168 (Metabolite of Deleobuvir)
Description: Area under the concentration-time curve of the analyte in plasma (CD 6168) over the time interval from 0 extrapolated to infinity. The descriptive statistics of the arms "Japanese 1200mg" and "Chinese 400mg" cannot be determined. The reason was that there were too few data to derive a terminal elimination rate constant (slope) to calculate AUC0-∞.
Time Frame: as for outcome 4
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol*h/L
Arm/Group | Caucasian 1200 mg | Japanese 400 mg | Japanese 800 mg | Chinese 800 mg | Chinese 1200 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
µmol*h/L | 15.8 (125.0) | 4.48 (85.8) | 11.0 (55.3) | 12.0 (25.1) | 22.2 (38.9)

10. Secondary Outcome: Tmax of CD 6168 (Metabolite of Deleobuvir)
Description: Time from dosing to the maximum measured concentration of the analyte in plasma (CD 6168).
Time Frame: as for outcome 4
Population: The PK analysis set.
Measure: Median (Full Range); unit: h
Arm/Group | Caucasian 1200 mg | Japanese 400 mg | Japanese 800 mg | Japanese 1200 mg | Chinese 400 mg | Chinese 800 mg | Chinese 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6
h | 6.01 [5.00 to 8.00] | 7.00 [5.00 to 8.00] | 6.00 [4.00 to 8.00] | 9.98 [5.07 to 10.00] | 6.00 [5.02 to 8.00] | 5.50 [5.00 to 8.00] | 7.00 [5.00 to 10.00]

11. Secondary Outcome: Cmax of CD 6168 (Metabolite of Deleobuvir)
Description: Maximum measured concentration of the analyte in plasma (CD 6168).
Time Frame: as for outcome 4
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol/L
Arm/Group | Caucasian 1200 mg | Japanese 400 mg | Japanese 800 mg | Japanese 1200 mg | Chinese 400 mg | Chinese 800 mg | Chinese 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6
µmol/L | 2.31 (80.7) | 0.57 (43.6) | 1.39 (34.3) | 2.65 (32.2) | 0.35 (109.0) | 1.66 (18.2) | 2.50 (30.9)

12. Secondary Outcome: AUC0-∞ of CD 6168 Acylglucuronide (Metabolite of Deleobuvir)
Description: Area under the concentration-time curve of the analyte in plasma (CD 6168 Acylglucuronide) over the time interval from 0 extrapolated to infinity. The descriptive statistics of the arms "Japanese 400mg", "Japanese 800mg", "Japanese 1200mg" and "Chinese 400mg" cannot be determined. The reason was that there were too few data to derive a terminal elimination rate constant (slope) to calculate AUC0-∞.
Time Frame: as for outcome 4
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol*h/L
Arm/Group | Caucasian 1200 mg | Chinese 800 mg | Chinese 1200 mg
Number analyzed (Participants) | 5 | 4 | 4
µmol*h/L | 1.27 (114) | 0.56 (17.5) | 1.01 (50.2)

13. Secondary Outcome: Tmax of CD 6168 Acylglucuronide (Metabolite of Deleobuvir)
Description: Time from dosing to the maximum measured concentration of the analyte in plasma (CD 6168 Acylglucuronide). The descriptive statistics of the arm "Chinese 400mg" cannot be determined due to limitation of available data above the "below limit of quantification (BLQ)".
Time Frame: as for outcome 4
Population: The PK analysis set.
Measure: Median (Full Range); unit: h
Arm/Group | Caucasian 1200 mg | Japanese 400 mg | Japanese 800 mg | Japanese 1200 mg | Chinese 800 mg | Chinese 1200 mg
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 6 | 6
h | 7.01 [5.00 to 8.00] | 8.00 [6.00 to 10.00] | 9.98 [6.00 to 10.00] | 10.00 [5.07 to 10.00] | 6.00 [5.00 to 8.00] | 8.00 [5.00 to 10.00]

14. Secondary Outcome: Cmax of CD 6168 Acylglucuronide (Metabolite of Deleobuvir)
Description: Maximum measured concentration of the analyte in plasma (CD 6168 Acylglucuronide).
  The descriptive statistics of the arm "Chinese 400mg" cannot be determined due to limitation of available data above the "below limit of quantification (BLQ)".
Time Frame: as for outcome 4
Population: The PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol/L
Arm/Group | Caucasian 1200 mg | Japanese 400 mg | Japanese 800 mg | Japanese 1200 mg | Chinese 800 mg | Chinese 1200 mg
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 6 | 6
µmol/L | 0.13 (62.3) | 0.03 (38.0) | 0.08 (48.2) | 0.11 (128.0) | 0.05 (29.0) | 0.07 (91.6)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed through the entire trial, from signing the informed consent (within 21 days before drug administration) onwards through the observational phase until the end-of-trial-examination (within 14 days after last trial procedure).
Description: Subjects were asked to spontaneously report any AEs as well as the time of onset, duration, and intensity. In addition, specific questions were asked whenever required or useful to more precisely describe an AE.
Groups:
- Placebo: All (Caucasian, Japanese and Chinese) subjects that received matching placebo. Oral with 240 mL of water in fed condition.
- 400 mg Deleobuvir: All (Japanese and Chinese) subjects that received 400 mg Deleobuvir. Oral with 240 mL of water in fed condition.
- 800 mg Deleobuvir: All (Japanese and Chinese) subjects that received 800 mg Deleobuvir. Oral with 240 mL of water in fed condition.
- 1200 mg Deleobuvir: All (Caucasian, Japanese and Chinese) subjects that received 1200 mg Deleobuvir. Oral with 240 mL of water in fed condition.
Arm/Group | Placebo | 400 mg Deleobuvir | 800 mg Deleobuvir | 1200 mg Deleobuvir
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12 | 0/12 | 0/18
Other Adverse Events (participants affected / at risk) | 5/14 | 1/12 | 2/12 | 14/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | 400 mg Deleobuvir (N=12) | 800 mg Deleobuvir (N=12) | 1200 mg Deleobuvir (N=18)
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 9
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 4
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 2 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.